CLINICAL TRIAL: NCT04054583
Title: The Impact of Renovations in Long Term Care Living Spaces on Residents With Dementia, Their Families and the Staff That Care for Them
Brief Title: Impact of Renovations in Long Term Care Living Spaces on Residents With Dementia, Their Families and Staff
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Riverview Health Centre Foundation (Other); Mitacs (Industry)
Responsible Party: Principal Investigator, Michelle Porter, Professor, University of Manitoba
Other Study IDs: E2016:084
Record Dates: First submitted 2019-07-22; First posted 2019-08-13 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Dementia
Keywords: Long-term care; Renovations; Residents; Family; Staff
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Residents: Residents living on a special care unit in a long-term care facility. All 60 residents residing in the unit pre- and post-renovation will be eligible, and all will have intermediate or advanced dementia.
  Interventions: Other: Renovation of long-term residential care living spaces
- Family Members: Family members are defined as the key person who supports the resident on a regular basis. This could include a spouse, adult child, adult grandchild, niece or nephew, close friend, former neighbour, or other significant person to the resident.
  Interventions: Other: Renovation of long-term residential care living spaces
- Staff: Staff are the people who work on the special care unit. They may work only briefly or work on the design of the renovations. Types include: managers, nurses, health care aides, recreation facilitators, social worker, occupational therapist, physiotherapist, rehabilitation assistant, speech language pathologist, physicians, designers, and cleaning staff.
  Interventions: Other: Renovation of long-term residential care living spaces

INTERVENTIONS:
Other: Renovation of long-term residential care living spaces — Living spaces of the long term care facility will be renovated.

SUMMARY:
A long-term care facility in central Canada planned to renovate their existing dementia care units. The overarching objective of this study was to examine the effects of the renovations on residents, family, and staff.

DETAILED DESCRIPTION:
A long-term care facility in central Canada renovated their existing dementia care units, which accommodates 60 residents with intermediate and advanced stages of dementia. The primary features of the renovation include physical upgrades and the addition of a large u-shaped activity pavilion. The overarching objective of this study was to examine the effects of these design transformations in the facility and grounds on residents, family, and staff. The overall project addressed the following questions:

* How does the long-term care unit renovation affect the health outcomes, quality of life, and lived experiences of residents?
* What are the effects of the long-term care unit renovation on care staff and family members?
* What aspects of the transformation were responsible for observed changes? And what aspects worked or did not?

A multi-component, mixed-methods (qualitative and quantitative) research plan was used in this project. Personal (resident, families, staff) and environmental variables (social interactions, implementation and use of technology and physical space) were assessed pre-renovation (spring/summer 2017) and post-renovation (summer 2019 and 2020). Due to the COVID-19 pandemic, plans for additional data collection in the summer of 2020 were not completed. With this mixed-methods research plan, the investigators gained valuable information about the renovation that is important for long term care facilities.

ELIGIBILITY:
Resident Inclusion Criteria:

* Currently living on special care unit for residents with intermediate to advanced dementia or cognitive impairment in a long-term care facility

Family Member Inclusion:

* Must have a family member/friend/neighbour currently living on the special care unit.
* For the QUALID, the family member must have visited the resident at least three out of the last seven days

Family Member Exclusion Criteria:

* Must be able to participate in-person.
* Must be able to communicate in English.
* Must be cognitively able to participate.

Staff Inclusion Criteria:

* Must currently work on the special care unit (either full or part-time or occasional)
* For the survey, staff must be able to read and understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents living on a special care unit for residents with intermediate to advanced dementia or cognitive impairment, their family members, and staff who care for them
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Satisfaction of Space on Resident Quality of Life and Family Interactions from Pre- to Post-renovation from Family Perspective Using Photovoice and Photo Elicitation | Perspectives taken a pre- and post-renovation (approximately 2 years later or whenever renovations are complete).
  Family member's perspective regarding whether the renovations have had an effect on the resident's quality of life and the quality of their family's interactions with the resident. This will be gathered using photovoice (participant taken photos) and photo elicitation (researcher taken photos). In this method, both photo types will be discussed in one interview at pre- and one interview at post-renovation to gather impressions of the space and its impact on resident quality of life and family interactions. This is a qualitative research method. It will assess impressions at pre-renovations and at post-renovations.
Changes in Space Utilization | Data will be collected for six months prior to and six months after the renovations (approximately 2 years later or whenever renovations are complete)
  Using a floor plan/map, observers will indicate the locations of occupants with a dot on a map and an activity code that indicates the behaviour of that person. Observations will occur every hour over 18 hours and over 6 days. This will show how the space is used before and after renovations.
Changes in Building Occupant Satisfaction Survey of Staff | Perspectives taken pre- and post-renovation (approximately 2 years later or whenever renovations are complete).
  Staff perspective of how the space is used and functions before and after renovations. This survey measures variables such as overall environmental satisfaction, including satisfaction with acoustics, lighting, indoor air quality, and thermal comfort. Participants are also asked to provide descriptions of personal workspace, window proximity and workstation tenure, job satisfaction and demand, and method of working/time allocation. This survey has demonstrated reliability (Cronbach's alpha=0.728 to 0.873) and validity when compared with physical environment measures. There are no sub-scales. Each question will be evaluated independently.

SECONDARY OUTCOMES:
Neuropsychiatric Symptoms of Residents from Six Months Prior to Renovation to Six Months Post-Renovation | Measures will be collected six months prior to renovations and and six months after renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Frequency of aggression or agitation as recorded in resident charts.
Physical Restraints of Residents from Six Months Prior to Renovation to Six Months Post-Renovation | Measures will be collected six months prior to renovations and and six months after renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Frequency of use of physical restraints as recorded in resident charts.
Anti-psychotic Medications and Sedatives with Residents from Six Months Prior to Renovation to Six Months Post-Renovation | Measures will be collected six months prior to renovations and and six months after renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Frequency of prescription of anti-psychotic medications and sedatives as recorded in resident charts.
Patient Safety Indicators of Residents from Six Months Prior to Renovations to Six Months Post-renovation: Frequency of medication errors and residents falls | Measures will be collected six months prior to renovations and six months after renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Frequency of medication errors and residents falls as recorded in administrative records.
Functional and Health Status of Residents: Changes in Sleep Records | Measures will be collected six months prior to renovations and six months after renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Using the Resident Assessment Inventory - Minimum Data Set 2.0 (RAI-MDS) data, the frequency of sleep record will be compared six months prior to the renovations and six months after renovations have been completed. Each resident's sleep status is recorded on an hourly basis throughout the night. RAI-MDS is a standardized measurement tool that is used in long term care facilities across Canada.
Functional and Health Status of Residents: Changes in Aggressive Behaviour Scale Scores | Measures will be collected six months prior to renovations and six months after renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Using the Resident Assessment Inventory - Minimum Data Set 2.0 (RAI-MDS) data, final scores of the Aggressive Behaviour Scale (ABS) will be compared six months prior to the renovations and six months after renovations have been completed. Behaviour items used to calculate the ABS are: verbally abusive, physically abusive, socially inappropriate/disruptive behaviour, and resists care. Indicators of behavioural symptoms are recorded as part of the MDS assessments and are based upon the frequency of the behaviour within the last 7 days. The outcome scores range from 0-12 which are indicative of the following aggressive behaviour categories: 0=non, 1-2=moderate, 3-5=severe, and 6-12=very severe. RAI-MDS is a standardized measurement tool that is used in long term care facilities across Canada.
Functional and Health Status of Residents: Changes in Cognitive Performance Scale Scores | Measures will be collected six months prior to renovations and six months after renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Using the Resident Assessment Inventory - Minimum Data Set 2.0 (RAI-MDS) data, final scores of the Cognitive Performance Scale (CPS) will be compared six months prior to the renovations and six months after renovations have been completed. The CPS is based on a predictive algorithm validated against the Mini-Mental State Examination. Scores of this scale range from 0 to 6, and identify the resident's level of impairment for the following 5 elements: comatose, short-term memory, cognitive skills for daily decision-making, making self understood, and eating. A higher score indicates increased impairment in cognitive function. RAI-MDS is a standardized measurement tool that is used in long term care facilities across Canada.
Functional and Health Status of Residents: Change in Pain Scale Scores | Measures will be collected six months prior to renovations and six months after renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Using the Resident Assessment Inventory - Minimum Data Set 2.0 (RAI-MDS) data, final scores of the Pain Scale will be compared six months prior to the renovations and six months after renovations have been completed. This was developed to examine the prevalence of pain experienced by residents in nursing homes. It has been validated against the Visual Analogue Scale and has been shown to be valid in detecting pain. Scores range 0-3 with higher scores indicating a more severe pain experience. RAI-MDS is a standardized measurement tool that is used in long term care facilities across Canada.
Functional and Health Status of Residents: Changes in Falls Risks Assessment Scale Scores | Measures will be collected six months prior to renovations and six months after renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Using the Resident Assessment Inventory - Minimum Data Set 2.0 (RAI-MDS) data, final scores of the Falls Risks Assessment Scale will be compared six months prior to the renovations and six months after renovations have been completed. RAI-MDS is a standardized measurement tool that is used in long term care facilities across Canada.
Functional and Health Status of Residents: Changes in the Index of Social Engagement Scale | Measures will be collected six months prior to renovations and six months after renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Using the Resident Assessment Inventory - Minimum Data Set 2.0 (RAI-MDS) data, final scores of the Index of Social Engagement Scale will be compared six months prior to the renovations and six months after renovations have been completed. Scores range 0-6 with higher scores indicating a higher level of social engagement. RAI-MDS is a standardized measurement tool that is used in long term care facilities across Canada.
Functional and Health Status of Residents: Changes in Resident's Engagement Level using the Pool Activity Level (PAL) tool | Measures will be collected six months prior to renovations and six months after renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Using the Resident Assessment Inventory - Minimum Data Set 2.0 (RAI-MDS) data, final scores of the PAL Tool will be compared six months prior to the renovations and six months after renovations have been completed. THE PAL Tool determines the person's current level of engagement and includes 4 activity levels: planned, exploratory, sensory, reflex. The PAL Checklist covers nine everyday activities: bathing/washing; getting dressed; eating; contact with others; group work skills; communication skills; practical activities (for example: craft, domestic chores, gardening); use of objects; and looking at a newspaper/magazine. Four descriptive statements are provided for each activity. The caregiver ticks the one that most accurately describes the individual's performance of that activity over the preceding two weeks. The number of statements selected for each level is totaled and the highest 'scoring' one indicates the individual's activity level.
Functional and Health Status of Residents: Changes in Depression Rating Scale Scores | Measures will be collected six months prior to renovations and six months after renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Using the Resident Assessment Inventory - Minimum Data Set 2.0 (RAI-MDS) data, final scores of the Index of Depression Rating Scale will be compared six months prior to the renovations and six months after renovations have been completed. This scale suggests possible clinical depression warranting further investigation. Scores range 0-14 with a score of 3 or more may indicate a potential or actual problem with depressions. RAI-MDS is a standardized measurement tool that is used in long term care facilities across Canada.
Functional and Health Status of Residents: Changes in Activities of Daily Living Self-Performance Hierarchy Scale Scores | Measures will be collected six months prior to renovations and six months after renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Using the Resident Assessment Inventory - Minimum Data Set 2.0 (RAI-MDS) data, final score of the Activities of Daily Living (ADL) Self-performance Hierarchy Scale will be compared six months prior to the renovations and six months after renovations have been completed. This scale reflects the disablement process by grouping ADL performance levels into discrete stages of loss (this is, early loss: personal hygiene; middle loss: toileting and locomotion; late loss: eating). Scores range 0-6 with higher scores indicating greater decline (progressive loss) in ADL performance. RAI-MDS is a standardized measurement tool that is used in long term care facilities across Canada.
Functional and Health Status of Residents: Changes in Activities of Daily Living Short Form Scale Scores | Measures will be collected six months prior to renovations and six months after renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Using the Resident Assessment Inventory - Minimum Data Set 2.0 (RAI-MDS) data, final scores of the Activities of Daily Living (ADL) Short Form Scale will be compared six months prior to the renovations and six months after renovations have been completed. This scale provides a measure of the resident's ADL self-performance status based on items that reflect stages of loss (early, middle and late loss). Scores range 0-16 with higher scores indicating more impairment of self-sufficiency in ADL Performance. RAI-MDS is a standardized measurement tool that is used in long term care facilities across Canada.
Functional and Health Status of Residents: Changes in Activities of Daily Living Long Form Scale Scores | Measures will be collected six months prior to renovations and six months after renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Using the Resident Assessment Inventory - Minimum Data Set 2.0 (RAI-MDS) data, final scores of the Activities of Daily Living (ADL) Long Form Scale will be compared six months prior to the renovations and six months after renovations have been completed. This scale provides measure of the resident's ability to perform ADLs. The ADL Long Form is more sensitive to clinical changes than the other ADL scales. Scores range from 0-28 with higher scores indicating more impairment of self-sufficiency in ADL performance. RAI-MDS is a standardized measurement tool that is used in long term care facilities across Canada.
Changes in Staffing from Pre- to Post-renovation: Worker's Compensation Board Claims | Data will be collected for six months prior to and six months after the renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Aggregated human resources data will be gathered of the number and type of worker's compensation board claims of staff working on the special care unit from pre- to post-renovation.
Changes in Staffing from Pre- to Post-renovation: Absenteeism | Data will be collected for six months prior to and six months after the renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Aggregated human resources data will be gathered of the total number of hours and average number of hours when staff have been absent from work due to illness from pre- to post-renovation
Changes in Staffing from Pre- to Post-renovation: Leave of Absence | Data will be collected for six months prior to and six months after the renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Aggregated human resources data will be gathered of the total number of hours staff have taken a leave of absence for any reason from pre- to post-renovation.
Changes in Staffing from Pre- to Post-renovation: Staff Retention | Data will be collected for six months prior to and six months after the renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Aggregated human resources data will be gathered on the total number of staff who worked on the special care unit prior to the renovations and were still working on the unit at post-renovation.
Changes in Staffing from Pre- to Post-renovation: Staff Turnover | Data will be collected for six months prior to and six months after the renovations have been completed (approximately 2 years later or whenever renovations are complete).
  Aggregated human resources data will be gathered on the total number of staff who worked on the special care unit prior to the renovations but were no longer working on the unit at post-renovation.
Changes in the Quality of Life in Late Stage Dementia (QUALID) Scores of Residents | Data will be taken pre- and post-renovation (approximately 2 years later or whenever renovations are complete). The QUALID takes approximately 10 minutes to complete whereas DCM occurs over 2 days.
  Quality of Life in Late stage Dementia (QUALID) questionnaire total score will be compared before and after renovations. The QUALID is completed by family who have visited a resident at least three of the last seven days. This is an 11-item interview that asks a family member or caregiver to rate how often a specific resident exhibits behaviours associated with quality of life (e.g., smiling, enjoying a meal). A 5-point scale captures the frequency of each item (total score ranging from 11 to 55). Lower scores reflected a higher quality of life (QOL). This interview takes 5-10 minutes to complete for each resident for whom we have consent/assent.
Changes in the Quality of Life of Residents: Dementia Care Mapping | Data will be taken pre- and post-renovation (approximately 2 years later or whenever renovations are complete). The QUALID takes approximately 10 minutes to complete whereas DCM occurs over 2 days.
  Dementia Care Mapping (DCM) involves observing residents over several hours. The goal of this assessment is to collect in-depth data regarding resident's behaviours and use of space/time during a discrete time period. Mapping takes place using a designated instrument by a certified mapper, and in communal care and living spaces. One to twenty four different domains are tracked that can be said to account for a high level or a low level of well-being or quality of life. Observations of family members may also occur for those who have provided consent. Observational data will be entered into a computer program that provides profiles of residents' mood, engagement and well-being. This provides a useful index of the relative well-being or detriments that affect an individual in a given space and given specific relational and care activities.
Use and Maintenance of Space from Pre- to Post-renovation | Perspectives taken pre- and post-renovation (approximately 2 years later or whenever renovations are complete).
  Key staff informants will participate in a walk-through interview where the informant and investigator walk through the unit and discuss the physical space. This is a qualitative interview.
Changes in Indoor Environment Measures: Dry Bulb Temperature | Data will be collected for prior to and after the renovations (approximately 2 years later or whenever renovations are complete)
  Measures will be taken of dry bulb temperature at pre- and post-renovations. Optimum comfort for sedentary work is between 20°C and 26°C, depending on the time of year and clothing worn.
Changes in Indoor Environment Measures: Air Speed | Data will be collected for prior to and after the renovations (approximately 2 years later or whenever renovations are complete)
  Measures will be taken of air speed at pre- and post-renovations. For an all air systems, air velocity (speed) should be typically 20 fpm (0.1m/sec) to 40 fpm (.2 m/sec) to be experienced by the occupant. 40 fpm would be experienced in a laboratory environment whereas 15-20 fpm would be typical for an office space.
Changes in Indoor Environment Measures: Relative Humidity | Data will be collected for prior to and after the renovations (approximately 2 years later or whenever renovations are complete)
  Measures will be taken of relative humidity at pre- and post-renovations. Indoor humidity level should be 30-50%. When outdoor temperature is below -10 degrees C, indoor relative humidity should be 30%.
Changes in Indoor Environment Measures: Light Level | Data will be collected for prior to and after the renovations (approximately 2 years later or whenever renovations are complete)
  Measures will be taken of light level at pre- and post-renovations. Light level should be a minimum 322.92 lux of continuous lighting levels in all corridors and enclosed stairways, bedrooms, vestibules, washrooms, and tub and shower rooms.
Changes in Indoor Environment Measures: Noise Level | Data will be collected for prior to and after the renovations (approximately 2 years later or whenever renovations are complete)
  Measures will be taken of noise level at pre- and post-renovations. Limit exposure to 85 decibels averaged over 8 hours, with a peak level of 140dB.
Changes in Indoor Environment Measures: Air Quality - Volatile Organic Compounds (VOC) | Data will be collected for prior to and after the renovations (approximately 2 years later or whenever renovations are complete)
  Measures will be taken of air quality based on concentrations of VOC at pre- and post-renovations. Recommended levels:
  Butadiene (1.7 µg/m3) Dichlorobenzene (60 µg/m3) Butoxyethanol 11000 µg/m3) Ethoxyethanol (70 µg/m3) Chloropropene (1 µg/m3)
Changes in Indoor Environment Measures: Air Quality - Carbon Dioxide (CO2) | Data will be collected for prior to and after the renovations (approximately 2 years later or whenever renovations are complete)
  Measures will be taken of air quality based on concentrations of CO2 at pre- and post-renovations. Exposure limits:
  * long-term exposure limit (24 hours): 11.5 mg/m3 (10 ppm)
  * short-term exposure limit (1 hour): 28.6 mg/m3 (25 ppm)
Changes in Indoor Environment Measures: Air Quality - Formaldehyde | Data will be collected for prior to and after the renovations (approximately 2 years later or whenever renovations are complete)
  Measures will be taken of air quality based on concentrations of formaldehyde at pre- and post-renovations. Exposure limits:
  * long-term exposure limit for 8 hours: 50 µg/m3 (40 ppb)
  * short-term exposure limit (1 hour): 123 µg/m3 (100 ppb)
Changes in Indoor Environment Measures: Air Quality - Airborne Particulates | Data will be collected for prior to and after the renovations (approximately 2 years later or whenever renovations are complete)
  Measures will be taken of air quality based on concentrations of airborne particulates at pre- and post-renovations.

OTHER OUTCOMES:
Process Evaluation | Prior to, during and after the renovation (approximately 2 years later or whenever renovations are complete)
  Documents (meeting minutes, training manuals, etc.) as well as staff interviews will be used to determine the context of units over the time of the renovation. For example, are there other changes occurring, beyond the renovation, that could have an effect on the residents, family and staff over the timeframe of the renovation project.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle M Porter, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No